CLINICAL TRIAL: NCT07354880
Title: Effect of Tirzepatide on Cardiovascular and Metabolic Parameters in Obese Adult Patients With Congenital Heart Disease
Acronym: TEACH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Katja Prokselj, Assoc. prof., senior consultant, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120-156/2025-2711-4
Record Dates: First submitted 2026-01-09; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight; Adult Congenital Heart Disease
Keywords: Obesity; adult congenital heart disease; tirzepatide; cardiovascular factors; metabolic factors
MeSH Terms: conditions — Obesity; Overweight; Heart Defects, Congenital | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trizepatide (Active Comparator): Tirzepatide (Munjaro), starting dose 2,5 mg subcutaneous weekly for 4 weeks, dosage increased monthly for 2.5 mg according to study protocol, based on clinical response and tolerability.
  Interventions: Drug: Treatment with tirzapatide
- Placebo (Placebo Comparator): Placebo 0.9% saline via identical pens administrated subcutaneous once weekly, same as active comparator, according to the same study protocol
  Interventions: Drug: Treatment with placebo

INTERVENTIONS:
Drug: Treatment with tirzapatide — Treatment with tirzepatide for 6 months, starting dosage 2,5 mg subcutaneous. Titration every 4 weeks by 2,5 mg increase, based on clinical response and tolerability of adverse effects, up to a maximum dose of 15 mg.
  Arms: Trizepatide
Drug: Treatment with placebo — Treatment with palcebo for 6 months, 0.9% saline via administrated via identical pens subcutaneous once weekly, same as active comparator, according to the same study protocol.
  Arms: Placebo

SUMMARY:
Several drugs have been shown effective in the treatment of obesity, with concomitant favourable cardiovascular effects. Today, there are no studies on novel anti-obesity drugs in patients with adult congenital heart disease (ACHD). Therefore, the investigators aim to study the effects of the anti-obesity drug tirzepatide (Munjaro) on cardiovascular and metabolic factors in obese patients with ACHD.

In a 24-week, randomized, open-label, placebo-controlled clinical trial the investigators will compare the effects of tirzepatide versus placebo in ACHD patients diagnosed with obesity. Patients will be randomized in a 1:1 ratio to either the intervention or placebo group. Participants will have monthly visits to monitor progress. At the beginning and end of the study, a full investigation protocol will be performed.

DETAILED DESCRIPTION:
Introduction Obesity is a complex multifactorial disease with major impact on the cardiovascular system and subsequent adverse cardiovascular events.

Congenital heart disease (CHD) is the most common congenital disease. With the advancement of the treatment nowadays around 90% of patients with mild, 75% with moderate, and 40% with complex congenital heart disease reach the age of 60 years. With aging, acquired heart disease is becoming more prevalent and poses a growing concern in adults with CHD (ACHD). The ACHD patients are at an increased risk for atherosclerotic cardiovascular disease and its risk factors. In comparison to the general population, patients with ACHD have more severe risk factors for atherosclerosis, which frequently clinically presents at an earlier age and has increased morbidity and mortality.

Among well known risk factors for atherosclerotic cardiovascular disease, obesity plays an important role. It is estimated that, similarly to general population, up to 40-50% of ACHD patients are overweight or obese. These patients are at an increased risk for arterial hypertension, hyperlipidaemia, and diabetes. The development of obesity in ACHD is multifactorial, potentially including inadequate education on healthy lifestyle, sedentary lifestyle, and overfeeding during infancy.

CHD is a long-life disease, requiring frequent interventions throughout life, among them also surgical and catheter interventions. Obesity poses a risk for complications in surgical and catheter interventions, which increase morbidity and mortality in these patients.

Novel pharmacological treatment of obesity is an emerging help in reducing not only weight in obese patients but also contributing to diminishing obesity-related adverse effects.

Tirzepatide (Mounjaro), a drug developed for the treatment of type 2 diabetes, is a dual glucose-dependent insulinotropic polypeptide and glucagon-like peptide-1 that has been recently approved also for the treatment of obesity. Studies have shown that treatment with tirzepatide significantly reduces blood pressure, LDL cholesterol, and triglycerides, all of them established cardiovascular risk factors. There is a large-scale ongoing study, assessing the impact of tirzepatide on major adverse cardiovascular events, such as myocardial infarction and stroke in patients with type 2 diabetes and cardiovascular disease. A recent study has shown that tirzepatide led to a lower risk of a composite of death from cardiovascular causes or worsening heart failure than placebo and improved health status in patients with heart failure with preserved ejection fraction and obesity.

Today, there are no studies on novel antiobesity drugs in patients with ACHD. Therefore, the investigators aim to study the effects of tirzepatide on cardiovascular and metabolic factors in obese patients with ACHD.

Aim of the study The investigators aim to determine the effects of the treatment with tirzepatide on obese patients with ACHD. The investigators will focus on several cardiovascular parameters, such as echocardiographic function of the left ventricle, exercise capacity parameters on exercise testing, blood pressure changes, changes in the arterial stiffness, and endothelial function. Metabolic parameters, encompassing weight change, blood sugar and lipid status, inflammation parameters, and hormones, will be assessed. The investigators expect that 24-week treatment with tirzepatide will result in the improvement of cardiovascular and metabolic parameters.

Study design The investigators designed a 24-week, randomized, open-label, placebo-controlled clinical trial to compare the effects of tirzepatide versus placebo in patients with ACHD diagnosed with obesity. Patients will be randomized in a 1:1 ratio to either the intervention or placebo group.

Study population and eligibility criteria The investigators will enroll approximately 30-40 participants with ACHD who meet the established criteria for pharmacological intervention in obesity, as outlined in current international guidelines. The cohort inclusion criteria will be limited to a body mass index (BMI) between 30 and 40 kg/m². To mitigate potential confounding variables, the study will exclude participants with secondary causes of obesity, such as thyroid disorders, autonomous glucocorticoid activity, or syndromic conditions. Additionally, any evident syndromic forms of obesity will be ruled out through clinical examination during the endocrinological assessment.

Patients with ACHD are followed in the tertiary national centre for ACHD at the Department of Cardiology, University Medical Centre Ljubljana. The patients will be enrolled during their regular follow-up at the outpatient clinic for ACHD. All potentially eligible patients will receive written and oral information about the study including the potential adverse effects of the treatment, the procedures conducted, the reporting of these effects, and the recommended measures upon their occurrence. A screening examination will be performed after the patient has agreed to participate and has signed the informed consent form. At the time of screening, the patients will undergo examinations to ensure that all inclusion criteria and none of the exclusion criteria are met. All patients who meet the inclusion and exclusion criteria at screening will be enrolled for randomization followed by a 24-week study period.

Intervention Tirzepatide (Mounjaro, Eli Lilly) will be administered as a subcutaneous injection using prefilled pens, following a modified titration protocol. Participants in the intervention group will begin with a 2.5 mg weekly dose for 4 weeks, followed by potential increases of 2.5 mg every 4 weeks, based on clinical response and tolerability of adverse effects, up to a maximum dose of 15 mg. Participants in the placebo group will receive 0.9% saline via identical pens. At the study's outset, participants will receive education on self-administration and perform their first injection under supervision in-clinic. Thereafter, participants will self-administer the treatment at home, attending monthly clinic visits for monitoring and dose adjustments.

Treatment allocation After the screening phase, participants will be randomized after the test day to one of the two study groups in a 1:1 ratio in accordance with a subject randomization list.

Trial visits and examinations The study will include two main sets of visits: an initial set before the start of treatment (V1) and a follow-up set after 24 weeks of treatment (V6). Throughout the treatment period, independent of the two main sets of visits (V1 and V6), participants will undergo monthly laboratory tests to monitor an extended panel of electrolytes, liver and kidney function tests to ensure safety (V2-5).

Visit 1 and 6 will include:

* Clinical examination
* Quality of life assessment, HADS, IPAQ, DEBQ, OP, FFQ and TFEQ-R18 questionnaire
* Heart rate and heart rate variability measurement
* Measurement of body composition, bone mineral density, and muscle strength
* Continuous glucose monitoring
* Basic and extended laboratory investigations
* Echocardiography
* Cardiopulmonary exercise testing
* Endothelial function and arterial stiffness measurement

Visit 2-5 will include:

* Clinical examination
* Basic laboratory investigations

ELIGIBILITY:
Inclusion Criteria:

* Obese or overweight adult patients with congenital heart disease
* BMI between 30 kg/m² and 40 kg/m²
* Prior comprehensive non-pharmacological and non-surgical management of obesity, including a history of at least 12 months of intensive lifestyle intervention with a maximum weight reduction of less than 5%
* Stable body weight within the three months preceding study enrollment (defined as weight fluctuations within 5%)
* No prior pharmacological or surgical interventions for obesity
* Euthyroid state
* Eumenorrhea or oligomenorrhea
* Ability to comprehend the study objectives and procedures
* Willingness to provide informed consent and to comply with the study protocol, including the use of highly effective contraception during the study period, with signed consent and agreement provided in duplicate
* Commitment to use highly reliable contraception and absence of plans for pregnancy within the 8 months following enrollment.

Exclusion Criteria:

* Down syndrome
* Type 2 diabetes
* Severe heart failure (NYHA IV), EF of systemic or subpulmonary ventricle < 30%, malignant arrhythmias, severe heart valve disease
* Personal history of malignancy, personal or family history of medullary thyroid carcinoma
* Personal history of pancreatitis or cholelithiasis
* Personal history of acute coronary events or hemodynamically significant coronary artery disease
* Current treatment with sympathomimetics or sympatholytic
* Psychiatric disorders, personal history of depressive disorders or suicidal ideation
* Pregnancy or lactation, postmenopausal, amenorrhea, reliance on natural contraception methods
* Excessive alcohol consumption
* Smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in exercise capacity after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  • Exercise capacity will be measured by maximum oxygen consumption at cardiopulmonary exercise testing, expressed in mL/kg/min.
Change in left ventricular systolic function after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Left ventricular systolic function will be evaluated echocardiographically by global longuitudinal strain (GLS), expressed in %
Change in cholesterol levels after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Patient's blood will be drawn between 8 and 9 am, after fasting. Cholesterol concentration will be expressed as mmol/L.

SECONDARY OUTCOMES:
Change in endothelial function after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Endothelial function will be measured by endothelium-dependent vasodilation, expressed in %.
Change in arterial stiffness after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Arterial stiffness ill be evaluated by pulse wave velocity, expressed in m/s.
Change in body weight after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Body weight will be measured in kilograms.

OTHER OUTCOMES:
Change of quality of life after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Quality of life will be evaluated by 36-Item Short Form Survey questionnaire and expressed on a scale scores, ranging from 0 to 100 (lower values representing worse outcome).
Change of anxiety and depression after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Anxiety and depression will be evaluated by Hospital Anxiety and Depression Scale questionnaire and expressed on a scale scores, ranging from 0 to 21 (lower values representing better outcome).
Change of physical activity after 6 months of treatment with tirzepatide. | From enrollment (visit 1) to the end of the treatment at 6 months (visit 6).
  Physical activity will be evaluated by International Physical Activity questionnaire and expressed in MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Janež, Prof., MD, PhD, Study Director — University Medical Centre Ljubljana, Slovenia; Margarita Brida, Ass. prof., MD, PhD, Study Chair — Royal Brompton Hospital, London, UK

IPD SHARING:
Plan to Share IPD: Yes
The data will be share in anonymized way, through publishing of manuscripts with study results.